CLINICAL TRIAL: NCT03053284
Title: Pasireotide for Prevention of Hypoglycemia in Patients With Hyperinsulinemic Hypoglycemia
Brief Title: Pasireotide in Hyperinsulinemic Hypoglycemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was withdrawn by Sponsor prior to start of study
Sponsor: Montefiore Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-7044
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Congenital Hyperinsulinism; Insulinoma; Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism; Insulinoma; Hyperinsulinism | interventions — pasireotide; Solutions; Injections; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Normal saline s.c. injection once
  Interventions: Drug: Saline Solution
- Pasireotide (Experimental): Pasireotide 0.6mg s.c. once
  Interventions: Drug: Pasireotide 0.6Mg Solution for Injection

INTERVENTIONS:
Drug: Pasireotide 0.6Mg Solution for Injection — Pasireotide 0.6Mg Solution for Injection will be given once per study visit
  Other Names: SOM230
  Arms: Pasireotide
Drug: Saline Solution — Saline Solution injection will be given once per study visit
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a small controlled pilot study to assess the effect of subcutaneous pasireotide on preventing hypoglycemia due to hyperinsulinism, including congenital hyperinsulinism and insulinoma.

DETAILED DESCRIPTION:
Pasireotide is a somatostatin analog with affinity for several somatostatin receptors including those on pancreatic beta cells; when activated these receptors affect the secretion of glucagon and insulin. Pasireotide is also known to decrease glucagon-like peptide 1 (GLP-1) and gastric inhibitory polypeptide (GIP) secretion. Hyperglycemia is a well-documented adverse effect of pasireotide in its approved indications for treatment of Cushing's disease and acromegaly.

In light of this, the investigators hypothesize that pasireotide may be an effective therapy for hypoglycemia due to hyperinsulinism. Therefore a small controlled pilot study to assess the effect of subcutaneous (s.c.) pasireotide on preventing hypoglycemia due to hyperinsulinism over 7 hours of observation in both fasting and fed states is proposed.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients aged 18 to 70 years old
2. Patients with hyperinsulinemic hypoglycemia due to either congenital hyperinsulinemic hypoglycemia or insulinoma, as determined by an endocrinologist
3. If no prior diagnosis of either insulinoma or congenital hyperinsulinemic hypoglycemia by an endocrinologist, the participant must meet the following criteria:

   * A history of symptoms of hypoglycemia, (with or without a blood glucose <50mg/dL at time of symptoms)
   * Improvement of symptoms with ingestion of carbohydrates
   * At least one documented blood glucose <50mg/dL with concomitant insulin >3 mmol/L and c-peptide >0.2nmol/L, with a negative sulfonylurea screen
   * At least 1 episode of glucose <50mg/dL in the last year
4. Written informed consent obtained prior to treatment to be consistent with local regulatory requirements
5. No evidence of significant liver disease:

   * Serum total bilirubin < 2 x ULN
   * INR < 1.3 unless on anticoagulation
   * ALT and AST < 2 x ULN
   * Alkaline phosphatase < 2.5 x ULN
6. Patients receiving anti-hypoglycemic treatment are eligible
7. Patients who are treatment naïve, or those who were previously, but not currently, treated with anti-hypoglycemic therapy are also eligible
8. Patients with insulinoma who are operative candidates are eligible if surgery is not emergently needed, and study participation would not delay the timing of a surgical intervention

Exclusion criteria:

1. Age <18, age >70 (for both insulinoma and congenital hyperinsulinism)
2. Known hypersensitivity to somatostatin or analogues
3. Diabetic patients with poor glycemic control as evidenced by HbA1c >8%
4. Patients who are hypothyroid and not on adequate replacement therapy
5. Patients with symptomatic cholelithiasis and acute or chronic pancreatitis
6. QTcF at screening > 450 msec in males and QTcF > 460 msec in females
7. Hypokalaemia, hypomagnesaemia, family history of long QT syndrome or concomitant medications with known risk of Torsades de pointes (TdP)
8. Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, advanced heart block, history of acute MI less than one year prior to study entry or clinically significant impairment in cardiovascular function
9. Severe non-malignant medical illness that may be jeopardized by treatment with a single dose of pasireotide
10. History of another primary malignancy, with the exception of locally excised non-melanoma skin cancer and carcinoma in situ of uterine cervix unless there is no evidence of disease in the last year
11. Patients with serum creatinine >2.0 X ULN
12. Patients with WBC <3 X 109/L; Hb 90% < LLN; PLT <100 X 109/L
13. Patients with the presence of active or suspected acute or chronic uncontrolled infection
14. Patients who have undergone major surgery/surgical therapy for any cause within 4 weeks prior screening
15. History of unexplained syncope or family history of idiopathic sudden death
16. Sexually active males unless they use a condom during intercourse while taking drug and for 3 months following last dose of pasireotide and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
17. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
18. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and 30 days following last dose of pasireotide.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemia | 7 hours
  Occurence, frequency and severity of hypoglycemia (serum glucose < 55 mg/dL)

SECONDARY OUTCOMES:
Serum glucose regulators | 7 hours
  Insulin, GLP-1, glucagon and cortisol levels

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 7 hours
  Collection of safety and adverse event data

CONTACTS AND LOCATIONS:
Overall Officials: Erika Brutsaert, M.D., M.P.H., Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmid HA, Brueggen J. Effects of somatostatin analogs on glucose homeostasis in rats. J Endocrinol. 2012 Jan;212(1):49-60. doi: 10.1530/JOE-11-0224. Epub 2011 Oct 10. PMID 21987782
- [Background] Braun M. The somatostatin receptor in human pancreatic beta-cells. Vitam Horm. 2014;95:165-93. doi: 10.1016/B978-0-12-800174-5.00007-7. PMID 24559918
- [Background] Boscaro M, Ludlam WH, Atkinson B, Glusman JE, Petersenn S, Reincke M, Snyder P, Tabarin A, Biller BM, Findling J, Melmed S, Darby CH, Hu K, Wang Y, Freda PU, Grossman AB, Frohman LA, Bertherat J. Treatment of pituitary-dependent Cushing's disease with the multireceptor ligand somatostatin analog pasireotide (SOM230): a multicenter, phase II trial. J Clin Endocrinol Metab. 2009 Jan;94(1):115-22. doi: 10.1210/jc.2008-1008. Epub 2008 Oct 28. PMID 18957506
- [Background] Yorifuji T. Congenital hyperinsulinism: current status and future perspectives. Ann Pediatr Endocrinol Metab. 2014 Jun;19(2):57-68. doi: 10.6065/apem.2014.19.2.57. Epub 2014 Jun 30. PMID 25077087
- [Background] de Heide LJ, Laskewitz AJ, Apers JA. Treatment of severe postRYGB hyperinsulinemic hypoglycemia with pasireotide: a comparison with octreotide on insulin, glucagon, and GLP-1. Surg Obes Relat Dis. 2014 May-Jun;10(3):e31-3. doi: 10.1016/j.soard.2013.11.006. Epub 2013 Dec 4. No abstract available. PMID 24448101
- [Background] Quinn TJ, Yuan Z, Adem A, Geha R, Vrikshajanani C, Koba W, Fine E, Hughes DT, Schmid HA, Libutti SK. Pasireotide (SOM230) is effective for the treatment of pancreatic neuroendocrine tumors (PNETs) in a multiple endocrine neoplasia type 1 (MEN1) conditional knockout mouse model. Surgery. 2012 Dec;152(6):1068-77. doi: 10.1016/j.surg.2012.08.021. Epub 2012 Oct 24. PMID 23102680
- [Background] Tirosh A, Stemmer SM, Solomonov E, Elnekave E, Saeger W, Ravkin Y, Nir K, Talmor Y, Shimon I. Pasireotide for malignant insulinoma. Hormones (Athens). 2016 Apr;15(2):271-276. doi: 10.14310/horm.2002.1639. PMID 26732164
- [Background] Eigler T, Ben-Shlomo A. Somatostatin system: molecular mechanisms regulating anterior pituitary hormones. J Mol Endocrinol. 2014 Aug;53(1):R1-19. doi: 10.1530/JME-14-0034. Epub 2014 Apr 29. PMID 24780840
- [Background] Hansen L, Hartmann B, Mineo H, Holst JJ. Glucagon-like peptide-1 secretion is influenced by perfusate glucose concentration and by a feedback mechanism involving somatostatin in isolated perfused porcine ileum. Regul Pept. 2004 Apr 15;118(1-2):11-8. doi: 10.1016/j.regpep.2003.10.021. PMID 14759551